CLINICAL TRIAL: NCT01173159
Title: Compassionate Use of a Fish Oil-derived Intravenous Fat Emulsion (Omegaven) to Reverse Parenteral Nutrition (PN) Induced Cholestasis
Brief Title: Compassionate Use of Omegaven to Reverse Parenteral Nutrition Induced Cholestasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-2314
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Results first posted 2020-05-08 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Cholestasis
Keywords: Parenteral Nutrition; Cholestasis
MeSH Terms: conditions — Cholestasis; Hyperphagia | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omegaven (Experimental): Subjects will receive Omegaven at a dose of up to 1 g/kg body weight/day until they no longer require Total Parenteral Nutrition or until their conjugated/direct bilirubin has normalized and their enteral lipid intake is sufficient to discontinue intravenous lipids.
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — For the first two days of treatment, subjects will receive Omegaven® at 0.5 g/kg per day to assess tolerance and will progress to a maintenance dosage of up to 1g/kg per day over 12 hours at an infusion rate of 1 g/kg/12 hours (10 ml/kg/12 hours). Dosing is based on previously described dosing of fish-oil emulsions as monotherapy noted within the literature. Omegaven® will be infused intravenously through either a central or peripheral catheter in conjunction with other parenteral nutrition containing dextrose and amino acids. Omegaven® is isotonic. It is compatible with parenteral nutrition solutions and may be co-infused via y-site.

SUMMARY:
The purpose of this research study is to see if giving Omegaven (an intravenous fat emulsion containing fish oil) instead of the current lipid emulsion, which contains fat derived from soybeans, as part of your child's intravenous (IV) nutrition therapy may be tolerated better. It may reduce the harmful effects to the liver, may stop any further liver damage and may reverse damage already done to the liver because of the prolonged use of nutrition through your child's IV.

DETAILED DESCRIPTION:
Enrollment of subjects into this study will occur for up to 4 years. Subjects will receive Omegaven at a dose of up to 1 g/kg body weight/day until they no longer require total parenteral nutrition or until their conjugated/direct bilirubin has normalized and their enteral lipid intake is sufficient to discontinue intravenous lipids.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages one month of age to 18 years of age
* Patients with intestinal failure on TPN
* Patients who have a conjugated/direct bilirubin of ≥3 mg/dl for more than weeks and in whom other causes of cholestasis have been excluded with reasonable certainty utilizing biochemical, serologic, microbiologic, and radiographic techniques. Liver biopsy is not required to rule out other disorders, but may be utilized at the clinician's discretion
* Patients in whom reduction of IV soy-based lipid to an average <1.2g/kg body weight/day has failed to reduce the conjugated/direct bilirubin within ≥ 30 days of implementation
* Willing to use birth control during study participation for females of child- bearing potential, as determined by investigator.
* Signed informed consent for use of Omegaven® obtained

Exclusion Criteria:

* Any of the contraindications to use of Omegaven®

  * Impaired lipid metabolism (triglycerides >1000 mg/dL) while on

    1g/kg/day or less of Intralipid
  * History of severe hemorrhagic disorders (ie. hemophilia, Von Willebrand disease, etc.)
  * Unstable diabetes mellitus
  * Collapse and shock
  * Stroke/ Embolism
  * Cardiac infarction within the last 3 months
  * Undefined coma status
  * Pregnancy (positive pregnancy test) prior to enrollment in the study for females of child-bearing potential
  * Females of child-bearing potential who are unwilling to use birth control during study participation
* Parental decision to forego the use of Omegaven®
* Known fish or egg allergy
* Pregnancy
* Causes of liver disease other than Parenteral Nutrition Associated Cholestasis

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Kocoshis, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omegaven
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Omegaven: Subjects will receive Omegaven at a dose of up to 1 g/kg body weight/day until they no longer require TPN or until their conjugated/direct bilirubin has normalized and their enteral lipid intake is sufficient to discontinue intravenous lipids.
  Omegaven: For the first two days of treatment, subjects will receive Omegaven® at 0.5 g/kg per day to assess tolerance and will progress to a maintenance dosage of up to 1g/kg per day over 12 hours at an infusion rate of 1 g/kg/12 hours (10 ml/kg/12 hours). Dosing is based on previously described dosing of fish-oil emulsions as monotherapy noted within the literature. Omegaven® will be infused intravenously through either a central or peripheral catheter in conjunction with other parenteral nutrition containing dextrose and amino acids. Omegaven® is isotonic. It is compatible with parenteral nutrition solutions and may be co-infused via y-site.
Arm/Group | Omegaven
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: months] | 6 [1 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change in Conjugated/Direct Bilirubin
Description: Change in conjugated/direct bilirubin level to below 1 mg/dl.
Time Frame: Completion of Therapy (time frame from 1-14 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 10
Participants | 4

2. Secondary Outcome: Number of Participants With a Change in Unconjugated/Total Bilirubin
Description: Change in unconjugated/total bilirubin level to below 1.1 mg/dL. General outcomes of participants are reported due to the enrollment of very few patients so that we have too small a cohort with which to assess achievement of our stipulated outcomes.
Time Frame: Completion of Therapy (time frame from 1-14 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 10
Participants | 5

3. Secondary Outcome: Number of Participants With a Change in Aspartate Transaminase (AST)
Description: Change in aspartate transaminase (AST) 57 units/L. General outcomes of participants are reported due to the enrollment of very few patients so that we have too small a cohort with which to assess achievement of our stipulated outcomes.
Time Frame: Completion of Therapy (time frame from 1-14 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 10
Participants | 2

4. Secondary Outcome: Number of Participants With a Change in Liver Enzyme (ALT)
Description: Change in liver enzyme ALT to below 59 unit/L. General outcomes of participants are reported due to the enrollment of very few patients so that we have too small a cohort with which to assess achievement of our stipulated outcomes.
Time Frame: Completion of Therapy (time frame from 1-14 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 10
Participants | 1

5. Secondary Outcome: Number of Participants With a Change in Liver Enzyme Alkaline Phosphatase
Description: Change in liver enzyme alkaline phosphatase to below 345 unit/L. General outcomes of participants are reported due to the enrollment of very few patients so that we have too small a cohort with which to assess achievement of our stipulated outcomes.
Time Frame: Completion of Therapy (time frame from 1-14 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 10
Participants | 3

6. Secondary Outcome: Number of Participants With a Change in Liver Enzyme Gamma-glutamyltransferase (GGT)
Description: Change in Liver Enzyme Gamma-glutamyltransferase (GGT) to below 15 unit/L. General outcomes of participants are reported due to the enrollment of very few patients so that we have too small a cohort with which to assess achievement of our stipulated outcomes.
Time Frame: Completion of Therapy (time frame from 1-14 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 10
Participants | 0

7. Secondary Outcome: Number of Participants With a Change in Triglycerides
Description: Change in Triglycerides to below 119 mg/dL. General outcomes of participants are reported due to the enrollment of very few patients so that we have too small a cohort with which to assess achievement of our stipulated outcomes.
Time Frame: Completion of Therapy (time frame from 1-14 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 10
Participants | 8

ADVERSE EVENTS:
Time Frame: 1 to 14 weeks of therapy
Arm/Group | Omegaven
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omegaven (N=10)
Sepsis (Blood and lymphatic system disorders) | 1 (2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Compartment Syndrome Following Surgery (Injury, poisoning and procedural complications) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Hyperkalemia Causing Cardiac Dysrhythmia (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Multisystem Organ Dysfunction related to IPEX (Congenital, familial and genetic disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omegaven (N=10)
Vomiting (General disorders) | 2 (3)
Fever (General disorders) | 3 (6)
Upper Respiratory Infection (General disorders) | 1 (1)
Phosporus Decreased (Investigations) | 1 (1)
Skin Irritation and breakdown (Skin and subcutaneous tissue disorders) | 2 (2)
Diaper Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary Vein Stenosis (Vascular disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal Fistula (Gastrointestinal disorders) | 2 (2)
Blood in Stool (Gastrointestinal disorders) | 1 (1)
Edema (Blood and lymphatic system disorders) | 2 (2)
Portal Hypertension (Gastrointestinal disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (2)
Irritability (General disorders) | 1 (1)
Dried blood near Anus (General disorders) | 1 (1)
Tachycardia and Tachypnea (Cardiac disorders) | 1 (1)
Culture Positive from Tracheostomy (Infections and infestations) | 1 (1)
Triglycerides Increased (Blood and lymphatic system disorders) | 1 (1)
Gull bladder sludge with intrahepatice biliary ductal dilation (Hepatobiliary disorders) | 1 (1)
Activated Partial Throboplastin Time Prolonged (Blood and lymphatic system disorders) | 1 (1)
Lethargy (General disorders) | 1 (2)
Platelet Count Decreased (Blood and lymphatic system disorders) | 1 (1)
Nasal Congestion (General disorders) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (General disorders) | 1 (1)
Decreased Respiratory Rate (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bleeding from nose (Hepatobiliary disorders) | 1 (1)
Abnormal CBC Differential with Active Bleeding (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
We enrolled very few patients so that we have too small a cohort with which to assess achievement of our outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT01173159/Prot_SAP_000.pdf